CLINICAL TRIAL: NCT02514551
Title: Randomized Phase 2 Trial Evaluating Alternative Ramucirumab Doses in Combination With Paclitaxel in Second-Line Metastatic or Locally Advanced, Unresectable Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: A Study of Ramucirumab (LY3009806) in Combination With Paclitaxel in Participants With Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15541; I4T-MC-JVCZ (Other: Eli Lilly and Company); 2014-005067-32 (EudraCT Number)
Record Dates: First submitted 2015-07-31; First posted 2015-08-03 (Estimated); Results first posted 2018-12-19 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06-01

CONDITIONS: Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma
Keywords: stomach cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Ramucirumab; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 12mg/kg Ramucirumab + 80 mg/m² Paclitaxel (Experimental): 12 milligram per kilogram (mg/kg) ramucirumab administered intravenously (IV) on day 1 and day 15 (28 day cycles) in combination with 80 milligram per square meter (mg/m²) paclitaxel administered IV on day 1, day 8 and day 15.
  Interventions: Drug: Ramucirumab; Drug: Paclitaxel
- 8 mg/kg Ramucirumab + 80 mg/m² Paclitaxel (Active Comparator): 8 mg/kg ramucirumab administered IV on day 1 and day 15 (28 day cycles) in combination with 80 mg/m² paclitaxel administered IV on day 1, day 8 and day 15.
  Interventions: Drug: Ramucirumab; Drug: Paclitaxel

INTERVENTIONS:
Drug: Ramucirumab — Administered IV
  Other Names: LY3009806; IMC-1121B; Cyramza
Drug: Paclitaxel — Administered IV

SUMMARY:
The main purpose of this study is to evaluate the efficacy of an alternative dose of ramucirumab in combination with paclitaxel in participants with second-line metastatic or locally advanced, unresectable gastric or gastroesophageal junction adenocarcinoma (GEJ).

ELIGIBILITY:
Inclusion Criteria:

* The participant has a diagnosis of gastric or GEJ adenocarcinoma.
* The participant has disease progression during or within 4 months after last dose of first-line chemotherapy or during or within 6 months after the last dose of neoadjuvant or adjuvant therapy.
* The participant received combination chemotherapy, which must include a platinum and/or a fluoropyrimidine and must not include a taxane or antiangiogenic agent.
* The disease is evaluable by imaging per Response Evaluation Criteria in Solid Tumors 1.1.
* The participant has an Eastern Cooperative Oncology Group performance status of 0 or 1.
* The participant has adequate organ function:

  * Total bilirubin ≤1.5 × the upper limit of normal (ULN) and alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3 × ULN. If the liver has tumor involvement, AST and ALT <5 × ULN.
  * Serum creatinine ≤1.5 × ULN or calculated creatinine clearance ≥50 milliliters/minute.
  * Urinary protein is <2+.
  * Absolute neutrophil count ≥1.5 × 10^9/liter (L), platelets ≥100 × 10^9/L, and hemoglobin ≥9 grams/deciliter (5.58 millimoles/L).
  * International normalized ratio ≤1.5 × ULN and partial thromboplastin time ≤5 seconds above ULN.
* The participant has an estimated life expectancy of minimum 12 weeks.
* The participant has resolution to Grade 1 or less by Common Terminology Criteria for Adverse Events Version 4.0, of all clinically significant toxic effects of previous therapy.
* The participant, if male, is sterile or agrees to use a reliable method of birth control.
* The participant, if female, is surgically sterile, is postmenopausal, or agrees to use a highly effective method of birth control.
* The participant, if female and of child-bearing potential, must have a negative pregnancy test.

Exclusion Criteria:

* The participant is receiving therapy with any of the following:

  * Nonsteroidal anti-inflammatory agents.
  * Other anti-platelet agents; Aspirin use at doses up to 325 milligrams (mg)/day is permitted.
* The participant received radiotherapy within 14 days prior to randomization.
* The participant received previous chemotherapy with a cumulative dose of >900 mg per meter squared (mg/m^2) of epirubicin or >400 mg/m^2 of doxorubicin.
* The participant has documented brain metastases or leptomeningeal disease.
* The participant has a significant bleeding disorder or vasculitis.
* The participant experienced any arterial thromboembolic event within 6 months.
* The participant has symptomatic congestive heart failure or symptomatic cardiac arrhythmia.
* The participant has uncontrolled hypertension, despite antihypertensive intervention.
* The participant underwent major surgery within 28 days.
* The participant has a history of gastrointestinal perforation or fistula within 6 months.
* The participant has a history of inflammatory bowel disease or Crohn's disease requiring medical intervention within 12 months.
* The participant has bowel obstruction or history of chronic diarrhea that is considered clinically significant.
* The participant has either of the following:

  * Child-pugh B or C cirrhosis.
* The participant has a serious illness or medical condition including:

  * Human immunodeficiency virus infection.
* The participant has a concurrent active malignancy other than the following:

  * Nonmelanomatous skin cancer.
  * In situ carcinoma of the cervix or other noninvasive carcinoma or in situ neoplasm.
* The participant has a serious nonhealing: (a) wound, (b) peptic ulcer, or (c) bone fracture.
* The participant experienced any Grade 3 or 4 venous thromboembolic event that is not adequately treated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2015-10-12 (Actual); Primary Completion 2017-10-27 (Actual); Study Completion 2018-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (49):
- United States (7):
  - City of Hope National Medical Center, Duarte, California
  - University of Kansas Medical Center, Westwood, Kansas
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Weill Cornell Medical College, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Scott & White Memorial Hospital & Clinic, Temple, Texas
  - Vista Oncology Inc. PS, Olympia, Washington
- Belgium (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brussels
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kortrijk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Namur
- Canada (2):
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Calgary
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Oshawa
- Czechia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brno
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nový Jičín
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prague
- Germany (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Frankfurt am Main
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ravensburg
- Greece (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Athens
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Haidari
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heraklion
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., N. Efkarpia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pátrai
- Italy (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cagliari
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cremona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Faenza
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Reggio Emilia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Giovanni Rotondo
- Spain (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Girona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Málaga
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santander
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seville
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valencia
- Sweden (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gothenburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Linköping
- Turkey (Türkiye) (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ankara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edirne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Istanbul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kayseri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Malatya
- Ukraine (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dnipropetrovsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kyiv
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lutsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sumy
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vinnitsa

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: Click here for more information about this study: A Study of Ramucirumab (LY3009806) in Combination With Paclitaxel in Participants With Gastric Cancer — http://www.lillytrialguide.com/EN-us/studies/cancer/jvcz

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Completers are defined as participants who died or had progressive disease (PD) or completed treatment or did not complete treatment and were followed for survival data. Final study data will be provided after study completion.
Period: Overall Study
Arm/Group | 12mg/kg Ramucirumab + 80 mg/m² Paclitaxel | 8 mg/kg Ramucirumab + 80 mg/m² Paclitaxel
Started | 123 | 122
Received at Least One Dose of Study Drug | 123 | 120
Completed | 123 | 119
Not Completed | 0 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Participant Never Treated | 0 | 2

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- 12mg/kg Ramucirumab + 80 mg/m² Paclitaxel: 12mg/kg ramucirumab administered intravenously (IV) on day 1 and day 15 (28 day cycles) in combination with 80 mg/m² paclitaxel administered IV on day 1, day 8 and day 15.
- Total: Total of all reporting groups
Arm/Group | 12mg/kg Ramucirumab + 80 mg/m² Paclitaxel | 8 mg/kg Ramucirumab + 80 mg/m² Paclitaxel | Total
Number analyzed (Participants) | 123 | 122 | 245
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (11.4) | 57.9 (12.3) | 58.3 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 44 | 84
  Male | 83 | 78 | 161
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 7 | 15
  Not Hispanic or Latino | 110 | 108 | 218
  Unknown or Not Reported | 5 | 7 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 119 | 117 | 236
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Greece | 10 | 11 | 21
  Canada | 0 | 4 | 4
  Sweden | 1 | 1 | 2
  Turkey | 24 | 16 | 40
  Belgium | 6 | 5 | 11
  United States | 16 | 8 | 24
  Czechia | 7 | 9 | 16
  Ukraine | 18 | 26 | 44
  Italy | 16 | 7 | 23
  Germany | 2 | 2 | 4
  Spain | 23 | 33 | 56

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) in Ramucirumab 12mg/kg Arm I4T-MC-JVCZ
Description: PFS was defined as time from the date of randomization(RD) to date of radiographic documentation of progression(RDP) or the date of death due to any cause, whichever is earlier as defined by RECIST v.1.1. Participants with no tumor progression and no death were censored at date of last adequate radiological assessment (AST) or date of RD(whichever is later).PD is at least a 20% increase in sum of diameters of target lesions,taking as reference the smallest sum on study.In addition to the relative increase of 20%,the sum must also demonstrate an absolute increase of at least 5 mm.The appearance of 1 or more new lesions is also considered progression.Non-Target PD is unequivocal progression of existing nontarget lesions.A participant with incomplete baseline disease had PFS time censored at the enrollment date.A participant not known to have died or have RDP as of the data inclusion cutoff date for the analysis had PFS time censored at date of the last complete RDP-free disease AST.
Time Frame: Randomization to Objective Progressive Disease or Death (Up To 21 Months)
Population: All randomized participants in arm 12mg/kg Ramucirumab + 80 mg/m² Paclitaxel. Number of participants censored: Ramucirumab 12 mg/kg + 80 mg/m² Paclitaxel= 25. All randomized participants (including the censored participants) were included in the analyses.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- I4T-MC-JVCZ: 12mg/kg Ramucirumab + 80 mg/m² Paclitaxel: 12mg/kg ramucirumab administered intravenously (IV) on day 1 and day 15 (28 day cycles) in combination with 80 mg/m² paclitaxel administered IV on day 1, day 8 and day 15.
Arm/Group | I4T-MC-JVCZ: 12mg/kg Ramucirumab + 80 mg/m² Paclitaxel
Number analyzed (Participants) | 123
months | 5.42 [4.40 to 6.01]
Statistical Analysis 1: Comparison: I4T-MC-JVCZ: 12mg/kg Ramucirumab + 80 mg/m² Paclitaxel; This analysis were comparison of PFS for participants treated with ramucirumab 12 mg/kg plus paclitaxel in Study I4T-MC-JVCZ versus placebo plus paclitaxel in I4T-IE-JVBE (NCT01170663) using meta-analysis. Placebo + 80 mg/m² Paclitaxel in I4T-IE-JVBE Number of participants: 335, Median (95% CI), months: 2.86 (2.79 to 3.02); Test type: Superiority; Hazard Ratio (HR) = 0.617, 95% CI 2-sided [0.447 to 0.853] — Unstratified cox proportional hazards model comparing Ramucirumab I4T-MC-JVCZ and I4T-IE-JVBE (NCT01170663)

2. Secondary Outcome: Progression Free Survival (PFS) Ramucirumab 12mg/kg Arm and 8mg/kg Arm in I4T-MC-JVCZ
Description: PFS was defined as time from the date of randomization(RD) to date of radiographic documentation of progression(RDP) or the date of death due to any cause, whichever is earlier as defined by RECIST v.1.1. Participants with no tumor progression and no death were censored at date of last adequate radiological assessment(AST) or date of RD(whichever is later).PD is at least a 20% increase in sum of diameters of target lesions,taking as reference the smallest sum on study.In addition to the relative increase of 20%,the sum must also demonstrate an absolute increase of at least 5 mm.The appearance of 1 or more new lesions is also considered progression.Non-Target PD is unequivocal progression of existing nontarget lesions.A participant with incomplete baseline disease had PFS time censored at the enrollment date.A participant not known to have died or have RDP as of the data inclusion cutoff date for the analysis had PFS time censored at date of the last complete RDP-free disease AST.
Time Frame: Randomization to Objective Progressive Disease or Death (Up To 21 Months)
Population: All randomized participants. Number of participants censored: Ramucirumab 12 mg/kg + Paclitaxel 80 mg/m2= 25 and 8 mg/kg Ramucirumab + 80 mg/m² Paclitaxel =23. All randomized participants (including the censored participants) were included in the analyses.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 12mg/kg Ramucirumab + 80 mg/m² Paclitaxel | 8 mg/kg Ramucirumab + 80 mg/m² Paclitaxel
Number analyzed (Participants) | 123 | 122
months | 5.42 [4.40 to 6.01] | 5.16 [3.81 to 5.65]
Statistical Analysis 1: Comparison: 12mg/kg Ramucirumab + 80 mg/m² Paclitaxel vs 8 mg/kg Ramucirumab + 80 mg/m² Paclitaxel; Test type: Superiority; Hazard Ratio (HR) = 0.963, 95% CI 2-sided [0.727 to 1.274] — Unstratified cox proportional hazards model

3. Secondary Outcome: Pharmacokinetics (PK): Minimum Concentration (Cmin) of Ramucirumab in Combination With Paclitaxel
Description: Pharmacokinetics (PK): Minimum Concentration (Cmin) of Ramucirumab in Combination with Paclitaxel
Time Frame: Cycle(C) 1 Day(D) 1: Prior to Infusion(PTI),1 to 1.5 hours(hrs) after end of Infusion(EOI); C1 D15: 3 days PTI; C2 D1: 3 days PTI; C2 D15: 3 days PTI,1 to 1.5 hrs after EOI; C3 D1 and 15: 3 days PTI; C4 D1: 3 days PTI and 1 to 1.5 hrs after EOI
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter (µg/mL)
Arm/Group | 12mg/kg Ramucirumab + 80 mg/m² Paclitaxel | 8 mg/kg Ramucirumab + 80 mg/m² Paclitaxel
Number analyzed (Participants) | 103 | 95
Microgram per milliliter (µg/mL)
  Cycle 1 Day 15 (Week 2) | 39.2 (43) | 21.4 (58)
  Cycle 2 Day 1 (Week 4): number analyzed (Participants) | 97 | 85
  Cycle 2 Day 1 (Week 4) | 63.6 (40) | 37.1 (50)
  Cycle 2 Day 15 (Week 6): number analyzed (Participants) | 84 | 69
  Cycle 2 Day 15 (Week 6) | 76.7 (42) | 43.5 (53)
  Cycle 3 Day 1(Week 8): number analyzed (Participants) | 74 | 58
  Cycle 3 Day 1(Week 8) | 91.2 (40) | 51.5 (55)
  Cycle 3 Day 15 (Week 10): number analyzed (Participants) | 62 | 57
  Cycle 3 Day 15 (Week 10) | 99.0 (44) | 52.9 (56)
  Cycle 4 Day 1 (Week 12): number analyzed (Participants) | 51 | 50
  Cycle 4 Day 1 (Week 12) | 101 (55) | 56.1 (56)

4. Secondary Outcome: Percentage of Participants Who Achieve Best Overall Tumor Response of Complete Response (CR) or Partial Response (PR) (Objective Response Rates [ORR])
Description: ORR was defined as the percentage of participants who achieved a PR or CR per RECIST v.1.1.CR is the disappearance of all target lesions.Any pathological lymph nodes(whether target or non-target)must have reduction in short axis to<10mm.Tumor marker results must have normalized.PR is at least a 30% decrease in the sum of diameter of target lesions,taking as reference the baseline sum diameters.ORR is calculated as a total number of participants with CR or PR divided by the total number of participants treated multiplied by 100.
Time Frame: Baseline to Objective Progressive Disease (Up To 21 Months)
Population: All randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | 12mg/kg Ramucirumab + 80 mg/m² Paclitaxel | 8 mg/kg Ramucirumab + 80 mg/m² Paclitaxel
Number analyzed (Participants) | 123 | 122
percentage of participants | 27.6 | 25.4

5. Secondary Outcome: Percentage of Participants Who Exhibit Stable Disease (SD) or Confirmed Response (CR) or Partial Response (PR) [Disease Control Rate (DCR)]
Description: DCR is defined as the percentage of participants who achieved CR, PR, or SD per RECIST v.1.1. CR is the disappearance of all target lesions. Any pathological lymph nodes (target or non-target) must have reduction in short axis to <10 mm.Tumor marker results must have normalized. PR is at least a 30% decrease in the sum of diameter of target lesions, taking as reference the baseline sum diameters. SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. PD is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.The appearance of 1 or more new lesions is also considered progression. Non-Target PD is unequivocal progression of existing nontarget lesions. DCR=CR+PR+SD/total number of participants*100.
Time Frame: Baseline to Objective Progressive Disease (Up To 21 Months)
Population: All randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | 12mg/kg Ramucirumab + 80 mg/m² Paclitaxel | 8 mg/kg Ramucirumab + 80 mg/m² Paclitaxel
Number analyzed (Participants) | 123 | 122
percentage of participants | 78.9 | 75.4

6. Secondary Outcome: Number of Participants With Anti-Ramucirumab Antibodies
Description: Participants who had anti-ramucirumab antibodies at postbaseline.
Time Frame: Cycle 1 Predose through Follow-up (Up To 24 Months)
Population: All randomized participants who received at least one dose of study drug and were evaluable for ramucirumab anti-drug antibody.
Measure: Count of Participants; unit: Participants
Arm/Group | 12mg/kg Ramucirumab + 80 mg/m² Paclitaxel | 8 mg/kg Ramucirumab + 80 mg/m² Paclitaxel
Number analyzed (Participants) | 105 | 89
Participants | 2 | 1

ADVERSE EVENTS:
Time Frame: Up To 40 Months
Description: All randomized participants who received at least one dose of study drug.
Arm/Group | 12mg/kg Ramucirumab + 80 mg/m² Paclitaxel | 8 mg/kg Ramucirumab + 80 mg/m² Paclitaxel
All-Cause Mortality (participants affected / at risk) | 81/123 | 76/120
Serious Adverse Events (participants affected / at risk) | 47/123 | 32/120
Other Adverse Events (participants affected / at risk) | 117/123 | 115/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 12mg/kg Ramucirumab + 80 mg/m² Paclitaxel (N=123) | 8 mg/kg Ramucirumab + 80 mg/m² Paclitaxel (N=120)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 3 (3)
Bone marrow failure (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4) | 3 (3)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiovascular insufficiency (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (5) | 2 (2)
Ascites (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 3 (6) | 1 (1)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 2 (2)
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumoperitoneum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Tongue oedema (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1)
Asthenia (General disorders) | 2 (2) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1)
General physical health deterioration (General disorders) | 2 (2) | 0 (0)
Localised oedema (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1)
Oedema (General disorders) | 1 (1) | 0 (0)
Organ failure (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallbladder rupture (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis toxic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 2 (3) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Enteritis infectious (Infections and infestations) | 1 (1) | 0 (0)
Escherichia infection (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 2 (2) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (2)
Pneumonia necrotising (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 6 (6) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour perforation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (2) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Oedema genital (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 12mg/kg Ramucirumab + 80 mg/m² Paclitaxel (N=123) | 8 mg/kg Ramucirumab + 80 mg/m² Paclitaxel (N=120)
Anaemia (Blood and lymphatic system disorders) | 34 (72) | 39 (77)
Leukopenia (Blood and lymphatic system disorders) | 9 (44) | 9 (18)
Neutropenia (Blood and lymphatic system disorders) | 22 (78) | 24 (62)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (10) | 4 (5)
Abdominal distension (Gastrointestinal disorders) | 7 (9) | 6 (8)
Abdominal pain (Gastrointestinal disorders) | 20 (31) | 19 (22)
Abdominal pain upper (Gastrointestinal disorders) | 8 (13) | 12 (16)
Ascites (Gastrointestinal disorders) | 9 (11) | 5 (8)
Constipation (Gastrointestinal disorders) | 23 (33) | 21 (27)
Diarrhoea (Gastrointestinal disorders) | 31 (78) | 35 (65)
Dysphagia (Gastrointestinal disorders) | 11 (12) | 4 (4)
Nausea (Gastrointestinal disorders) | 27 (52) | 38 (95)
Stomatitis (Gastrointestinal disorders) | 15 (19) | 18 (41)
Vomiting (Gastrointestinal disorders) | 29 (51) | 27 (44)
Asthenia (General disorders) | 15 (35) | 19 (49)
Fatigue (General disorders) | 43 (85) | 46 (82)
Oedema peripheral (General disorders) | 10 (11) | 16 (22)
Pyrexia (General disorders) | 9 (10) | 8 (8)
Alanine aminotransferase increased (Investigations) | 14 (27) | 7 (8)
Aspartate aminotransferase increased (Investigations) | 20 (43) | 8 (15)
Blood alkaline phosphatase increased (Investigations) | 9 (25) | 10 (14)
Blood bilirubin increased (Investigations) | 8 (12) | 2 (3)
Neutrophil count decreased (Investigations) | 30 (91) | 24 (60)
Platelet count decreased (Investigations) | 9 (15) | 7 (13)
Weight decreased (Investigations) | 14 (16) | 13 (17)
White blood cell count decreased (Investigations) | 13 (33) | 14 (35)
Decreased appetite (Metabolism and nutrition disorders) | 25 (41) | 32 (58)
Hyperglycaemia (Metabolism and nutrition disorders) | 8 (18) | 11 (20)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 10 (13) | 14 (34)
Hyponatraemia (Metabolism and nutrition disorders) | 7 (13) | 7 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (13) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (13) | 9 (14)
Myalgia (Musculoskeletal and connective tissue disorders) | 11 (18) | 9 (16)
Dysgeusia (Nervous system disorders) | 5 (5) | 9 (13)
Headache (Nervous system disorders) | 10 (12) | 9 (12)
Neuropathy peripheral (Nervous system disorders) | 15 (38) | 15 (22)
Paraesthesia (Nervous system disorders) | 13 (30) | 13 (29)
Peripheral sensory neuropathy (Nervous system disorders) | 8 (15) | 20 (46)
Proteinuria (Renal and urinary disorders) | 9 (19) | 8 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (17) | 8 (11)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 11 (15) | 6 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 12 (13)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 26 (43) | 28 (36)
Alopecia (Skin and subcutaneous tissue disorders) | 19 (19) | 24 (28)
Hypertension (Vascular disorders) | 24 (44) | 21 (46)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2015-05-07): https://cdn.clinicaltrials.gov/large-docs/51/NCT02514551/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-15): https://cdn.clinicaltrials.gov/large-docs/51/NCT02514551/SAP_001.pdf